CLINICAL TRIAL: NCT00148122
Title: A Phase II Trial Evaluating Weekly Docetaxel and Capecitabine in Patients With Metastatic or Advanced, Locally, Recurrent Head and Neck Cancer
Brief Title: A Study of a New Combination and Schedule of Chemotherapy Drugs for the Treatment of Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Francis (Frank) Worden, Principal Investigator, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2-33; Legacy IRBMED 2002-747 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Head and Neck Cancer
Keywords: Squamous cell cancer of the oral cavity and pharynx
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Docetaxel (1000mg PO BID days 5-18 of each Cycle) and Capecitabine (30mg/m2/week IV days 1, 8, &15)
  Interventions: Drug: Docetaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Docetaxel — Each four-week cycle consists of three infusions through a vein of docetaxel, on days 1, 8, and 15. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule. If the subject's disease has not decreased significantly but there is no evidence the disease is getting worse, he/she will continue on the same treatment until: a) there is evidence that the treatment is no longer working to control the growth of his/her disease, b) He/she experiences unacceptable toxicity, c) his/her disease progresses, or d) he/she chooses to stop therapy.
  Other Names: US Brand Name: Taxotere
Drug: Capecitabine — Each four-week cycle consists of fourteen days of a medication that the subject will take two times a day orally, on days 5-18. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule. If the subject's disease has not decreased significantly but there is no evidence the disease is getting worse, he/she will continue on the same treatment until: a) there is evidence that the treatment is no longer working to control the growth of his/her disease, b) He/she experiences unacceptable toxicity, c) his/her disease progresses, or d) he/she chooses to stop therapy.
  Other Names: US Brand Name(s): Xeloda

SUMMARY:
The purpose of this study is to determine the effectiveness and side effects of a new combination and schedule of chemotherapy drugs in the treatment of head and neck cancer. Patients with advanced or recurrent head and neck cancer, which is untreatable by surgery or radiation therapy are eligible for this study. Standard treatment for advanced or recurrent head and neck cancer involves the use of chemotherapy.

DETAILED DESCRIPTION:
Approximately 28,900 patients will be diagnosed with squamous cell cancers of the oral cavity and pharynx in the year 2002. Of these, an estimated 7,400 patients will present with metastases or develop recurrent disease, which is not amenable to surgery or radiation therapy. Palliative chemotherapy is thus the only treatment option. Currently, combinations of cisplatin and 5-fluorouracil are used as first line treatment strategies, with median times to progression of 2.5 to 3 months and median survival rates of 5 to 7 months. The time to achieve maximum response with combination therapy is on average 4 months.

Taxanes, with their unique mechanism of microtubule stabilization, have demonstrated response rates similar to standard, first line combination regimens. Several phase II studies have evaluated the efficacy of single agent docetaxel in head and neck cancer patients. Cumulative response rates were approximately 30%, with higher response rates observed in patients receiving no prior chemotherapy. Docetaxel has also been used in combination with cisplatin and cisplatin and 5-fluorouracil. Although response rates with such combination regimens were superior to the use of single agent docetaxel, grade 3 and 4 toxicities were also more prevalent.

Capecitabine (Xeloda®), a fluoropyrimidine carbamate, is an oral prodrug, which is converted in tumor tissues to 5-fluorouracil through multienzymatic activation. Capecitabine (Xeloda®) has documented activity in breast and colorectal cancers and is widely administered. Because 5-fluorouracil has efficacy in the treatment of head and neck cancer, it is reasonable to consider that such tumors will respond to capecitabine. To date, there are no published trials using capecitabine (Xeloda®) in the treatment of metastatic head and neck cancer patients. However, clinical trials are ongoing in the U.S. and Europe with promising results.

In preclinical models, a synergistic interaction between capecitabine and docetaxel has been documented. One possible explanation for the synergy is that docetaxel up-regulates tumor levels of thymidine phosphorylase, the enzyme essential for the activation of capecitabine and 5'-dFUrd to 5-fluorouracil. Clinically, O'Shaughnessy, et al. recently reported improved survival with docetaxel/capecitabine combination therapy in patients with metastatic breast cancer, who previously failed anthracycline-containing chemotherapy. In this phase III study, patients were stratified according to previous exposure to paclitaxel and then randomized to capecitabine (Xeloda®) (1250 mg/m2 twice daily, days 1-14) plus docetaxel (75 mg/m2 day 1, repeated every 21 days) versus docetaxel alone. Grade 3 and 4 toxicities were more common in the docetaxel/capecitabine combination arm. Capecitabine (Xeloda®) and docetaxel were interrupted and the dosages reduced by 25% in patients who experienced a second occurrence of a given grade 2 toxicity, or any grade 3 toxicity, suggesting that the starting dosages were perhaps too high.

The role of chemotherapy in metastatic head and neck cancer is limited to palliation of the symptoms of disease. Platinum and 5-fluorouracil combinations remain standard first line treatment strategies. The taxanes have been shown to have similar efficacy to such first line regimens and are often used as salvage treatment for patients with metastatic disease. Given that docetaxel has documented clinical efficacy in head and neck cancer and that there are preclinical data to suggest synergy with docetaxel and capecitabine, it is reasonable to consider using these agents in combination to treat head and neck cancer patients. Moreover, capecitabine and docetaxel have distinct mechanisms of action and no overlap of key toxicities. A recent phase I/II study by Tonkin, et al. in metastatic breast cancer patients demonstrated activity and less toxicity when docetaxel 30 mg/m2/week (day 1 and 8 q21 days) was combined with capecitabine 1800 mg/m2/day (14 of 21 days). In another phase I study by Nadella, et al. weekly docetaxel (36 mg/m2 ) was combined with 14 days of capecitabine (up to 1500 mg/m2/day) over a course of 28 days. Antitumor responses were observed in patients with breast, colon, and bladder cancers. Hence, we propose this study whereby patients with previously treated, metastatic/recurrent head and neck cancer will receive treatment with docetaxel and capecitabine.

To reduce the potential for toxicity, we will use a modification of the Nadella regimen. Docetaxel will be administered weekly at a dosage of 30 mg/m2 for 3 out of every 4 weeks and capecitabine will be administered at a flat dosage of 2000 mg per day (1000 mg p.o. b.i.d.) for two weeks out of every 4 weeks. The justification for using a flat dosage of capecitabine versus a calculated dosage is based on pharmacokinetic data that show no change in clearance of capecitabine with changes in BSA. We plan to use a fixed dose of 2000 mg qd (1000 mg q am and 1000 mg q pm). Fixed dosing of capecitabine is convenient and feasible, as shown in a prior University of Michigan study in breast cancer patients. In another study Schott, et al. informally piloted the combination of weekly docetaxel 36 mg/m2 and 1500 mg twice daily (3000 mg/day) x 14 days capecitabine in metastatic breast cancer patients, and found it to be without unexpected or untoward side effects. Additionally, to take advantage of the time course of upregulation of TP in the preclinical models, the capecitabine dose will be given on days 5-18. In a flat dosing scheme, the Nadella regimen would have administered an average dose of 2125 mg qd for 14 days, assuming an average BSA of 1.7 m2. We plan to round this dosage downward to 2000 mg per day x 14 days; therefore, our regimen will use a slightly lower dosage of capecitabine. We feel that our proposed slightly lowered dose (closer to Nadella phase I dosing vs. Tonkin) of capecitabine is justified for the following reasons:

1. The Nadella study was performed in a group of patients with solid tumor malignancies that were refractory to conventional therapy or for whom no effective therapy existed. ECOG performance status (PS) was 1 or 2 in 5/17 (30%) patients, 10/17 patients had received 2 or more lines of previous chemotherapy, and 7/17 patients had received previous radiotherapy. Based on data from previous treatment of head and neck cancer patients at the University of Michigan, the patient population to be enrolled in this trial is expected to be 60% PS 0 and 40% PS 1, and some will have received prior chemotherapy and/or radiotherapy. Like the Nadella patient population, a majority of our patients have been pretreated and are of poorer health.
2. Dose interruptions and modifications are built into the protocol so that appropriate changes in treatment can be made in patients with Grade I or II toxicity, before the toxicity becomes Grade III or greater. Since the docetaxel is given weekly, and the capecitabine is administered daily, if patients are experiencing toxicity within a cycle, the dose of either can be held or modified.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented advanced, locally recurrent, or metastatic head and neck carcinoma, which is untreatable by surgical resection or radiation therapy.
* Prior chemotherapy for advanced/metastatic disease is allowed (1 regimen only).
* Patients must be taxane-naïve (no prior docetaxel or paclitaxel).
* Patients who have received chemoradiation as a primary therapy for advanced head and neck cancer are eligible.
* Patients must have measurable or evaluable disease. Pre-study imaging for disease assessment must be done within 28 days of registration.
* Patients with brain metastases are eligible if they have been stable for at least six weeks post-radiation therapy.
* Aged 18 years or older
* Performance status of 0-2 by Zubrod criteria.
* Life expectancy of at least 12 weeks.
* Hematologic: absolute neutrophil count (ANC) equal to or > 1,500/mm3; hemoglobin equal to or > 8.0 g/dl; platelets equal to or > 100,000/mm3.
* Total bilirubin must be within normal institutional limits (WNL).
* Transaminases (AST/SGOT and ALT/SGPT) may be up to 2.5 X the institutional upper limit of normal (ULN) if alkaline phosphatase is less than ULN, or alkaline phosphatase may be up to 4 X ULN if transaminases are less than ULN.
* A calculated creatinine clearance of > 50 ml/min
* Women of childbearing potential must have a negative pregnancy test at baseline, prior to receiving any study drug. (Pregnant or lactating patients are excluded.)
* Patients of reproductive potential must practice effective contraception while on study and for at least six months after receiving the last dose of study drug.
* All patients must sign an informed consent prior to enrollment.
* No prior history of malignancy, except for adequately treated skin cancer or in situ cervical carcinoma or any other cancer in complete remission for at least two years.

Exclusion Criteria:

* Patients with congestive heart failure, second or third degree heart block or recent myocardial infarction within 12 months from registration are not eligible.
* Peripheral neuropathy equal to or greater than grade 2.
* Patients with a history of severe hypersensitivity reaction to drugs formulated with polysorbate 80.
* Use of standard chemotherapy or investigational agents for treatment of head and neck cancer within 28 days of 1st dose of study drug.
* Any medical or psychiatric illness which, in the opinion of the principal investigator, would compromise the patient's ability to tolerate this treatment regimen.
* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
* Pregnant or lactating women, women of childbearing potential with either a positive pregnancy test (PPT) at baseline, or sexually active females not using a reliable contraceptive method while on study and for at least six months after chemotherapy. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.)
* Sexually active patients not using a reliable contraceptive method while on study and for at least six months after chemotherapy.
* Patients with malabsorption syndromes will be excluded. Administration of capecitabine through feeding tubes is permitted.
* Serious concurrent infections.
* Any other serious uncontrolled medical or surgical conditions that the investigator feels might compromise study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-11; Primary Completion 2008-08 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Worden, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Capecitabine: Docetaxel (1000mg PO BID days 5-18 of each Cycle) and Capecitabine (30mg/m2/week IV days 1, 8, &15)
  Docetaxel: Each four-week cycle consists of three infusions through a vein of docetaxel, on days 1, 8, and 15. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule.
  Capecitabine: Each four-week cycle consists of fourteen days of a medication that the subject will take two times a day orally, on days 5-18. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule.
Period: Overall Study
Arm/Group | Docetaxel and Capecitabine
Started | 40
Completed | 38
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Although 40 patients were enrolled, 2 patients withdrew consent after treatment started, therefore only 38 were included in baseline analysis.
Groups:
- Arm 1: Docetaxel (1000mg PO BID days 5-18 of each Cycle) and Capecitabine (30mg/m2/week IV days 1, 8, &15)
  Docetaxel: Each four-week cycle consists of three infusions through a vein of docetaxel, on days 1, 8, and 15. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule.
  Capecitabine: Each four-week cycle consists of fourteen days of a medication that the subject will take two times a day orally, on days 5-18. If the subject's disease has decreased significantly, he/she will continue to receive docetaxel on the every four-week schedule.
Arm/Group | Arm 1
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 59.46 [39.86 to 75.08]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status score is an attempt to quantify a cancer patients' general well-being and activities of daily life. It runs from 0 to 5, with 0 denoting perfect health and 5 death
  participants
    0 (Asymptomatic) | 27
    1 (Symptomatic but Completely Ambulatory) | 9
    2 (Symtomatic; <50% in Bed During the Day) | 2
Histology [Number; unit: participants]
  Squamous Cell Cancer | 36
  Adenocarcinoma | 1
  Others | 1
Disease Extent [Number; unit: participants]
  Local Regional | 13
  Distant | 17
  Local Regional Distant | 7
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate at 4 Months
Description: Disease was assessed by radiologic imaging and RECIST (Response Evaluation Criteria in Solid Tumors) was used to determine response: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 4 months
Population: 40 patients were enrolled. 2 patients withdrew consent and 2 patients were not evaluable per protocol criteria: A patient will be considered evaluable for response if they received at least 2 cycles of chemotherapy, OR if they have obvious clinical signs of disease progression on physical examination after one cycle of chemotherapy.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 36
percentage of participants | 16

2. Secondary Outcome: Frequency of Grade III/IV Toxicities Experienced by Participants
Description: The frequency of grade 3 and grade 4 adverse events experienced by all treated participants.
Time Frame: 30 days post treatment
Population: 40 patients were enrolled. 2 patients withdrew consent, therefore only 38 were included in the toxicity analysis.
Measure: Number; unit: participants
Arm/Group | Arm 1
Number analyzed (Participants) | 38
participants
  Grade 3 and 4 Lymphopenia | 8
  Grade 3 and 4 Infection w/o Neutropenia | 5
  Grade 3 and 4 Fatigue | 4
  Grade 3 and 4 Leukocytes | 4
  Grade 3 and 4 Stomatitis | 4
  Grade 3 and 4 Neutrophils | 3
  Grade 3 and 4 Diarrhea | 2
  Grade 3 and 4 Hand-Foot Skin Reaction | 2
  Grade 3 and 4 Hemoglobin | 2
  Grade 3 and 4 Platelets | 2
  Grade 3 and 4 Allergic Reaction | 1
  Grade 3 and 4 Anorexia | 1
  Grade 3 and 4 Cardiac-Ischemia | 1
  Grade 3 and 4 Dysphagia | 1
  Grade 3 and 4 Dyspnea | 1
  Grade 3 and 4 Abnormal ENT Examination | 1
  Grade 3 and 4 Edema Limbs | 1
  Grade 3 and 4 Febrile Neutropenia | 1
  Grade 3 and 4 Hand-Foot Syndrome | 1
  Grade 3 and 4 Hyperglycemia | 1
  Grade 3 and 4 Hyponatremia | 1
  Grade 3 and 4 Infection with Unknown ANC | 1
  Grade 3 and 4 Infection, Lung | 1
  Grade 3 and 4 Melena | 1
  Grade 3 and 4 Mental Status Changes | 1
  Grade 3 and 4 Mucositis | 1
  Grade 3 and 4 Nausea | 1
  Grade 3 and 4 Oral Pain | 1
  Grade 3 and 4 Pain, Extremity | 1
  Grade 3 and 4 Pharyngolaryngeal Pain | 1
  Grade 3 and 4 AST Elevation | 1
  Grade 3 and 4 Vomiting | 1

3. Secondary Outcome: Probability of Progression Free Survival
Description: The estimated 1 year progression free survival. Progression was defined, using RECIST (Response Evaluation Criteria In Solid Tumors Criteria), as a 20% increase in the sum of the longest diameter of target lesions, the development of any new lesion, or the significant clinical deterioration related to the progression of patient's disease. The probability of progression-free survival was presented in a Kaplan-Meier curve to illustrate the distribution of progression time. The median time to progression was determined with a 95% CI (Confidence Interval).
Time Frame: 1 year post treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm 1
Number analyzed (Participants) | 36
percentage of patients | 25 [12.4 to 39.8]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for all patients up to 30 days post treatment.
Description: Although 40 patients were enrolled, 2 patients withdrew consent after treatment started, therefore only 38 were included in toxicity analysis.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 25/38
Other Adverse Events (participants affected / at risk) | 36/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=38)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
CNS hemorrhage/bleeding (Nervous system disorders) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Constitutional Symptoms-Other (General disorders) | 1 (1)
Diarrhea (no colostomy) (Gastrointestinal disorders) | 1 (1)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage-Other (Injury, poisoning and procedural complications) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 1 (1)
Infection, Lung (pneumonia) (Infections and infestations) | 1 (1)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (2)
Mental status changes (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy - motor (Nervous system disorders) | 1 (2)
Pain-Other (General disorders) | 1 (1)
Pericardial effusion/pericarditis (Cardiac disorders) | 1 (1)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin infection (Infections and infestations) | 1 (2)
Stomatitis/pharyngitis (Gastrointestinal disorders) | 1 (1)
Syndromes-Other (General disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vision-double vision (diplopia) (Eye disorders) | 1 (1)
Vital capacity decreased (Investigations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=38)
Abdominal pain or cramping (Gastrointestinal disorders) | 4 (6)
Alkaline phosphatase (Investigations) | 10 (19)
Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Auditory/Hearing-Other (Ear and labyrinth disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dehydration (Metabolism and nutrition disorders) | 7 (8)
Diarrhea (no colostomy) (Gastrointestinal disorders) | 11 (20)
Dizziness/lightheadedness (Nervous system disorders) | 6 (7)
Dysphagia, esophagitis, odynophagia (Gastrointestinal disorders) | 9 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (13)
Ear, nose and throat examination abnormal (Investigations) | 2 (3)
Edema (General disorders) | 8 (13)
Edema limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 22 (33)
Fever (General disorders) | 2 (4)
Hand-and-foot syndrome (General disorders) | 2 (5)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 5 (7)
Headache (Nervous system disorders) | 5 (6)
Hemoglobin (Investigations) | 20 (56)
Hemoglobin decreased (Investigations) | 6 (6)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hemorrhage-Other (Injury, poisoning and procedural complications) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (60)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (38)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (48)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 11 (19)
Hyponatremia (Metabolism and nutrition disorders) | 18 (27)
Hypotension (Vascular disorders) | 3 (3)
Infection without neutropenia (Infections and infestations) | 5 (5)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Leukocytes (total WBC) (Investigations) | 12 (33)
Leukopenia (Investigations) | 2 (2)
Lymphopenia (Investigations) | 18 (46)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 3 (3)
Mood alteration-depression (Psychiatric disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 16 (22)
Neuropathy - motor (Nervous system disorders) | 4 (4)
Neuropathy-sensory (Nervous system disorders) | 7 (9)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6 (8)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain-Other (General disorders) | 10 (15)
Palpitations (Cardiac disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Platelet count decreased (Investigations) | 3 (3)
Platelets (Investigations) | 6 (13)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Proctitis (Gastrointestinal disorders) | 2 (2)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3)
Rash/dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Rigors, chills (General disorders) | 2 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 12 (20)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 12 (18)
Salivary gland changes (Gastrointestinal disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3)
Stomatitis/pharyngitis (Gastrointestinal disorders) | 13 (19)
Tearing (watery eyes) (Eye disorders) | 3 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Voice changes/stridor/larynx (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 5 (6)
Weight loss (Metabolism and nutrition disorders) | 5 (5)
Wound-infectious (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No